CLINICAL TRIAL: NCT01808365
Title: Neisseria Meningitidis Carriage Study
Brief Title: N. Meningitidis Carriage Study
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114991
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Infections, Meningococcal
Keywords: Neisseria meningitidis; Philippines; carriage; meningococcus
MeSH Terms: conditions — Meningococcal Infections | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Throat swab

GROUPS / COHORTS (1):
- Study cohort
  Interventions: Procedure: Posterior pharyngeal swab; Other: Data collection

INTERVENTIONS:
Procedure: Posterior pharyngeal swab — Posterior pharyngeal swabs will be tested for the presence of N. meningitidis.
  Other Names: Throat swab
Other: Data collection — Collection of socio-demographic data and recording of serious adverse events by interview of subjects or subjects' parents/legally acceptable representatives.

SUMMARY:
This carriage study aims to evaluate the presence of meningococcus in Asian populations (and potential for disease) and explore the extent and serogroup distribution of meningococci circulating in the population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol or subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject/from the parent(s)/LAR of the subject.
* Asymptomatic subjects attending a school or university.
* A male or female between, and including 5 and 24 years of age at the time of enrollment.

Exclusion Criteria:

* Subjects who have received a meningococcal conjugate vaccine.
* Use of any investigational or non-registered product within one week before the enrollment visit.
* Acute respiratory tract infection within 14 days of sample collection.
* Immune deficiencies, haematological disorders and oncological disease.
* Use of steroids or immunosuppressant drugs within 14 days of sample collection.
* Administration of antibiotics within the 2 weeks preceding the collection of sample.
* Cranio-facial malformations prohibiting the collection of posterior pharyngeal swabs.
* Child in care.

Ages: 5 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy subjects aged between 5 and 24 years attending a school or university in the Philippines.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2013-08-02 (Actual); Primary Completion 2014-03-25 (Actual); Study Completion 2014-03-25 (Actual)

PRIMARY OUTCOMES:
Assessing the carriage prevalence of N.meningitidis using posterior pharyngeal swabs | At enrollment (Day 0)

SECONDARY OUTCOMES:
The serogroup (determined by Polymerase Chain Reaction) of any isolated N. Meningitidis colonies | At enrollment (Day 0)
Further characterization of any carried N. meningitidis using Multi Locus Sequence Typing | At enrollment (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Manila, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114991 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114991 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114991 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114991 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114991 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114991 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114991 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register